CLINICAL TRIAL: NCT01378923
Title: Pilot Evaluation of the Re-Entry Values and Mindfulness Program (REVAMP) With Jail Inmates
Brief Title: Evaluation of Re-Entry Values and Mindfulness Program (REVAMP) With Jail Inmates
Acronym: REVAMP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: George Mason University (Other)
Responsible Party: Principal Investigator, June Tangney, Professor, George Mason University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCT-01
Record Dates: First submitted 2011-06-17; First posted 2011-06-23 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Impulsive Behavior; Substance Abuse; HIV Risk Behavior; Anxiety; Depression; Criminogenic Thinking
Keywords: Mindfulness; Values; Jail Inmates; Impulsivity; Substance Abuse; HIV risk behavior; Anxiety; Depression; Criminogenic Thinking
MeSH Terms: conditions — Impulsive Behavior; Substance-Related Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Values-based mindfulness group (Experimental): The Re-entry values and mindfulness program (REVAMP) is an 8 session group intervention designed for jail inmates nearing release into the community
  Interventions: Behavioral: REVAMP
- Treatment as usual (Other): has access to standard jail interventions and programs
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: REVAMP — The Re-entry values and mindfulness program (REVAMP) is an 8 session group intervention designed for jail inmates nearing release into the community
  Arms: Values-based mindfulness group
Behavioral: TAU — have access to standard jail programs and services
  Arms: Treatment as usual

SUMMARY:
This is a pilot study to examine the acceptability and effectiveness of the Re-Entry Values and Mindfulness Program (REVAMP), a group intervention for jail inmates. It is hypothesized that REVAMP will reduce post-release recidivism, substance abuse, and HIV risk behavior.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Must be male
* Must be currently incarcerated jail inmate
* Must be sentenced
* Sentence must be short enough to serve out sentence at the Adult Detention Center
* Release date must follow projected final session of treatment
* Must speak, read, and write in English with sufficient proficiency to use workbook and participate in group sessions
* Must be assigned to the jail's "general population"

Exclusion Criteria:

* Actively psychotic
* Assigned "keep separate" from other group members

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Recidivism - Self Report of undetected crimes | 3 months post-release
Recidivism - Self Report of Arrests | 3 months post-release
Recidivism - Official Records of arrests | 3 months post-release
Substance Dependence symptoms - Texas Christian University (TCU) measure | 3 months post-release
HIV Risk Behavior - Sex and Intravenous Drug Use (IDU) - TCU | 3 months post-release
Acceptability - number of participants who report finding the treatment helpful and number who would recommend the treatment to a friend | 1 week post-treatment

SECONDARY OUTCOMES:
Mindfulness - Self report using Mindfulness Inventory: Nine Dimensions (MI:ND) | 1 week post-treatment and 3 months post-release
Self Control - Self report using Brief Self control Scale (BSC) | post-treatment and 3 months post-release
Self-Compassion - Self report using Neff's scale | 1 week post-treatment and 3 months post-release
Distress-Driven Impulsivity - Behavioral measure using Balloon Analog Reaction Test (BART) preceded by mirror tracing task | 1 week post-treatment
Psychological Symptoms - Self report using Personality Assessment Inventory | 1 week post-treatment and 3 months post-release

CONTACTS AND LOCATIONS:
Overall Officials: June P Tangney, PhD, Principal Investigator — George Mason University
Locations (1):
- Fairfax County Adult Detention Center, Fairfax, Virginia, United States